CLINICAL TRIAL: NCT05436769
Title: An Open Label, Randomized, Single Dose, Two-way Crossover , Two-Period, Two-Treatment, Two-Sequence Bioequivalence Study of Klaribact Tablet (Clarithromycin 500 mg), Compared With Reference Product, Klaricid Tablet (Clarithromycin 500 mg) in Healthy Adult Male Subjects
Brief Title: Bioequivalence Study of Klaribact (Clarithromycin) 500 mg, Film Coated Tablet
Acronym: BE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Karachi (Other)
Collaborators: Merck Pvt. Ltd, Pakistan (Unknown); Center for Bioequivalence Studies and Clinical Research (Other)
Responsible Party: Principal Investigator, Dr. Muhammad Raza Shah, Professor, University of Karachi
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CB-006-CLA-2012
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Healthy Volunteers; Bioequivalence Study
Keywords: Bioequivalence Study; Clarithromycin Tablet
MeSH Terms: interventions — Clarithromycin

STUDY DESIGN:
Intervention Model Description: A single center, open Label, Randomized, Two Way Cross over, Two Period, Two Treatment, two Sequence Bioequivalence Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Drug (Experimental): Klaribact (Clarithromycin 500 mg) Film Coated Tablet (Merck Pvt. Ltd, Pakistan)
  Interventions: Drug: Klaribact 500 mg Clarithromycin Tablet; Drug: Klaricid 500 mg Clarithromycin Tablet
- Reference Drug (Active Comparator): Klaricid 500 mg (Clarithromycin 500 mg) Film Coated Tablet (Abbot Laboratories (Pakistan) Limited)
  Interventions: Drug: Klaribact 500 mg Clarithromycin Tablet; Drug: Klaricid 500 mg Clarithromycin Tablet

INTERVENTIONS:
Drug: Klaribact 500 mg Clarithromycin Tablet — A single dose consisting of one Tablet of either test drug (Klaribact 500 mg) or reference drug (Klaricid 500mg) administered to each of the subjects in fasting condition with 240 mL water in both Periods alternatively.
Drug: Klaricid 500 mg Clarithromycin Tablet — A single dose consisting of one Tablet of either test drug (Klaribact 500 mg) or reference drug (Klaricid 500mg) administered to each of the subjects in fasting condition with 240 mL water in both Periods alternatively.

SUMMARY:
This is An Open Label, Randomized, Single Dose, Two Way Cross over, Two Period, Two Treatment, Two Sequence Bioequivalence Study to compare the rate and extent of absorption of Klaribact FC Tablet (Clarithromycin 500 mg) with Reference Product, Klaricid FC Tablet (Clarithromycin 500 mg) in healthy adult male subjects under fasting condition.

DETAILED DESCRIPTION:
The study will be conducted on 24 healthy adult male subjects in two Periods i.e. period I and II. The study subjects will stay at the clinical trial site for 35 hours, 11 hours before and 24 hours after the drug administration. All 24 subjects will be divided in two groups of 12 subjects in each group. One group will be treated with the test drug (T) and the other one with reference drug (R) in Period I. After the wash-out period of 7 days, the volunteers in these groups will receive the alternate treatment sequence (RT) in Period II.

Blood samples will be collected at 0 hr (before drug administration) 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8,10, 12, 16 and 24 hours after drug administration for quantification of Clarithromycin in plasma through LCMS/MS validated method.

ELIGIBILITY:
Inclusion Criteria:

* All subjects should be healthy and free from any epidemic, contagious or measurable disease (e.g. Malaria, Dengue).
* Age range for inclusion will be 18-50 year.
* BMI for all Subjects will be between 18.5-26.9 kg/m2.
* Participant capable of understanding the informed consent.
* Non Smokers, who have not smoked in last 3 months.
* Medical history, physical examination and screening tests must fall in normal range, unless the investigator considers the abnormality to be clinically not significant.
* Clinical laboratory test results should be within a normal range.
* Participants (who can read and understand urdu) should be able to give informed consent, understand and sign the Informed Consent Form.
* Participants should have adequate organ function (i.e., kidney, liver and heart).
* Subjects with negative urine screen for drugs of abuse. All subjects will have urine samples assayed for the presence of drugs of abuse as part of the clinical screening procedures and at each study period check-In.

Exclusion Criteria:

* Any active allergic disease or a history of any significant allergic disease (e.g. Rhinitis, dermatitis, asthma).
* Known hypersensitivity to Investigational drug(s).
* Abnormal results of blood and urine tests conducted at screening unless the investigator considers an abnormality to be clinically irrelevant.
* Presence or history of cardiac (e.g. Myocardial Infarction, arrythmia), renal (e.g.renal insufficiency) , hepatic (e.g. hepatic impairment) , organ insufficiency, bone marrow disease, hematological abnormality (e.g. leukemia, anemia),photosensitivity, neurological disorders (e.g. Alzheimer's disease) or gastrointestinal disease known to interfere with the drug absorption, distribution, metabolism or elimination (e.g. dysphagia).
* History or presence of any musculo skeletal disease (e.g. Tendonitis).
* Subject donated blood (450ml) within 12 weeks minimum preceding the study. 19
* Alcoholic or with a history of chronic alcohol intake or consumed alcohol or Gutka in last 3 months.
* Ingestion of OTC drug, within 14 days of drug administration (e.g. aspirin, ibuprofen).
* History of intake of any prescribed medicine (e.g. captopril, sumatriptan) during a period of 30 days, prior to drug administration day of study.
* Ingestion of investigational drug within 30 days, prior to investigational drug administration in the study.
* Ingestion of any known hepatic or renal clearance altering agents (e.g. erythromycin, cimetidine, barbiturates, phenothiazines, etc.) for a period of 30 days, prior to study initiation. Drug interaction section at 5.12 should be considered.
* Subjects with an uncontrolled medical condition (i.e., hypertension, cardiac arrhythmias, CHF) that places the patient at risk by participating in the study.
* Subjects with known HIV, hepatitis B or C infection or autoimmune diseases.
* History of drug exposure which, in the opinion of Investigator, amounts to drug abuse.
* Participation in other drug studies within three months prior to study initiation.
* Subjects with any physical/mental disability.
* Limited mental capacity to the extent that the subject is unable to provide legal consent and information regarding the side effects or tolerance of the study drug.
* Pregnancy or breast feeding, women of child bearing age who are not using a recognized form of contraception for at least last 30 days or using hormonal contraception, are also excluded.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-10-23 (Actual); Primary Completion 2012-11-02 (Actual); Study Completion 2012-12-25 (Actual)

PRIMARY OUTCOMES:
maximum plasma drug concentration | up to 24 hours post dose
  maximum drug concentration in plasma after dosing
AUC last (AUC 0-t) | 0 to 24 hours post dose
  Area under plasma concentration time curve from zero to time of the last measurable concentration
AUC total (AUC 0-∞) | 0 to 24 hours post dose
  area under the plasma concentration-time curve from zero to infinity.

SECONDARY OUTCOMES:
Time to reach maximum plasma concentration | up to 24 hours post dose
  Time required for the drug to reach maximum plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Muhammad R Shah, PhD, Principal Investigator — CBSCR, ICCBS, University of Karachi, Pakistan; Dr. Naghma Hashmi (Co-PI), PhD, Principal Investigator — CBSCR, ICCBS, University of Karachi, Pakistan
Locations (1):
- Center for Bioequivalence Studies and clinical research (CBSCR), ICCBS, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Un-identified individual participant data (IPD) will be available to other researchers on reasonable request to the principal investigator